CLINICAL TRIAL: NCT02159118
Title: A Trial of the Vidacare Powered Bone Marrow Aspiration and Core Biopsy System (OnControl by Vidacare) Compared to Traditional Manual Devices in Children
Brief Title: A Study Comparing Use of Manual and Power Bone Marrow Aspiration and Biopsy Devices in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Principal Investigator, Chatchawin Assanasen, MD, Associate Professor, Pediatric Hematology/Oncology, The University of Texas Health Science Center at San Antonio
Organization: Teleflex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2012
Record Dates: First submitted 2014-05-15; First posted 2014-06-09 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2014-08

CONDITIONS: Bone Marrow Aspiration and Biopsy Specimen Collection
Keywords: bone marrow aspiration; bone marrow biopsy; OnControl; powered bone marrow aspiration and biopsy device; standard manual bone marrow aspiration and biopsy device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual bone marrow aspiration and biopsy procedure (Active Comparator): Manual bone marrow aspiration and biopsy device
  Interventions: Device: Manual bone marrow aspiration and biopsy device
- Powered bone marrow aspiration and biopsy procedure (Active Comparator): Powered bone marrow aspiration and biopsy device
  Interventions: Device: Powered bone marrow aspiration and biopsy device

INTERVENTIONS:
Device: Manual bone marrow aspiration and biopsy device — Use of the manual bone marrow aspiration and biopsy device to collect bone marrow aspiration and bone marrow biopsy specimens.
  Arms: Manual bone marrow aspiration and biopsy procedure
Device: Powered bone marrow aspiration and biopsy device — Use of the powered bone marrow aspiration and biopsy device to collect bone marrow aspiration specimens and bone marrow biopsy specimens.
  Other Names: OnControl
  Arms: Powered bone marrow aspiration and biopsy procedure

SUMMARY:
The purpose of this study is to compare use of a powered bone marrow aspiration and biopsy device (OnControl) to use of a standard manual bone marrow aspiration and biopsy device to obtain bone marrow biopsy specimens in children. The hypothesis is that use of the powered device will improve the quantity and quality of bone marrow biopsy specimens when compared to the manual device.

DETAILED DESCRIPTION:
The purpose of this randomized, prospective trial is to compare use of the standard manual bone marrow aspiration and biopsy device to use of the powered bone marrow aspiration and biopsy device (OnControl) to obtain bone marrow biopsy specimens in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and assent for minors over the age of seven years must be obtained before any trial-related activities are initiated
* Patients requiring bone marrow aspirations and/or biopsies as part of standard diagnosis and treatment
* Treated at Christus Santa Rosa Children's hospital
* Age 2 to 18 years
* Male or female
* Supportive family with willingness to participate in completing questionnaires
* English or Spanish primary language

Exclusion Criteria:

* Patients who are pregnant
* Patients with hemorrhagic disorders such as congenital coagulation factor deficiencies disseminated intravascular coagulation and concomitant use of anticoagulants
* Patients with a skin infection or recent radiation therapy at the sampling site
* Patients with bone disorders such as osteomyelitis or osteogenesis imperfecta

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chatchawin Assanasen, MD, Principal Investigator — Christus Santa Rosa Children's Hospital
Locations (1):
- Christus Santa Rosa Children's Hospital, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Bone Marrow Aspiration and Biopsy Procedure: Manual bone marrow aspiration and biopsy device
  Manual bone marrow aspiration and biopsy device: Use of the manual bone marrow aspiration and biopsy device to collect one bone marrow aspiration and bone marrow biopsy specimen.
- Powered Bone Marrow Aspiration and Biopsy Procedure: Powered bone marrow aspiration and biopsy device
  Powered bone marrow aspiration and biopsy device: Use of the powered bone marrow aspiration and biopsy device to collect one bone marrow aspiration and bone marrow biopsy specimen.
Period: Overall Study
Arm/Group | Manual Bone Marrow Aspiration and Biopsy Procedure | Powered Bone Marrow Aspiration and Biopsy Procedure
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study were included in the baseline analysis, as the required sample size for the study was met. No participants were excluded from analysis. Analysis was made per protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Bone Marrow Aspiration and Biopsy Procedure | Powered Bone Marrow Aspiration and Biopsy Procedure | Total
Number analyzed (Participants) | 22 | 22 | 88
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 22 | 22 | 44
  (all) | 10 (5.3) | 9.7 (4.8) | 9.84 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 22 | 22 | 44
  Female | 8 | 10 | 18
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States: number analyzed (Participants) | 22 | 22 | 44
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percent of Hematopoietic Tissue Present in Bone Marrow Biopsy Specimens Obtained Using the Manual Device and Powered Device
Description: Bone marrow biopsy specimens will be evaluated by a blinded pathologist and measured for percent of hematopoietic tissue present. Higher percentage of hematopoietic tissue present in a biopsy specimen indicates a larger quantity of specimen for pathological evaluation.
Time Frame: within 24 hours of bone marrow sampling procedure
Population: All participants enrolled in the study were included in analysis, as the required sample size for the study was met. No subjects were excluded from analysis. Analysis was made per protocol.
Measure: Mean (Standard Deviation); unit: % Hematopoetic tissue present
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
% Hematopoetic tissue present | 42.5 (21.8) | 55.8 (19.4)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Bone Marrow Biopsy Specimen Size (Length) Obtained Using the Manual Device and the Powered Device
Description: bone marrow biopsy specimens will be evaluated by a blinded pathologist and measured for length.
Time Frame: within 24 hours of the bone marrow sampling procedure
Population: All participants enrolled in the study were included in the analysis, as the required sample size for the study was met. No participants were excluded from analysis. Analysis was made per protocol.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
mm | 13.9 (3.4) | 13.4 (4.7)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.65, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Bone Marrow Biopsy Specimen Size (Width) Obtained Using the Manual Device and the Powered Device
Description: bone marrow biopsy specimens will be evaluated by a blinded pathologist and measured for width.
Time Frame: within 24 hours of the bone marrow sampling procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
mm | 1.4 (0.3) | 1.8 (0.2)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Bone Marrow Biopsy Specimen Size (Volume) Obtained Using the Manual Device and the Powered Device
Description: bone marrow biopsy specimens will be evaluated by a blinded pathologist and measured for volume
Time Frame: within 24 hours of the bone marrow sampling procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
mm3 | 23.8 (11.5) | 36.5 (16.1)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Bone Marrow Biopsy Specimen Capture Rate for the Manual Device and the Powered Device
Description: number of needle passes required to capture one bone marrow biopsy specimen using the manual device and the powered device
Time Frame: at time of the bone marrow sampling procedure
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: needle passes
Units Other Than Participants: needle passes
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
Number analyzed (needle passes) | 24 | 31
needle passes | 1.1 (0.3) | 1.4 (0.7)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Amount of Time Lapsed From Needle to Skin Contact to Bone Marrow Aspiration Specimen Acquisition Using the Manual Device and the Powered Device
Description: measurement of the amount of time required to acquire a bone marrow aspiration specimen. timing starts when the bone marrow aspiration and biopsy needle first contacts the skin and ends when the aspiration specimen has been collected.
Time Frame: at time of the bone marrow sampling procedure
Population: All participants enrolled in the study were included in the analysis as the required sample size for the study was met. No participants were excluded from analysis. Analysis was made per protocol.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
seconds | 55 (34.1) | 53.2 (30.5)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Patient Level of Post-procedural Pain Following Use of the Manual Device and the Powered Device
Description: Within 4 hours of the bone marrow sampling procedure, the patient will report their level of pain post-procedure using the Wong-Baker FACES pain rating scale. The scale measures pain from 0-10, where higher numbers represent worse pain.
Time Frame: within 4 hours of the bone marrow sampling procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
units on a scale | 0.27 (0.94) | 0.68 (1.36)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Operator Satisfaction With Manual Device and Powered Device
Description: Device operators will report their level of satisfaction with use of the manual device and the powered device to perform the bone marrow sampling procedure. Level of satisfaction is reported using a 0 to 10 scale, where higher numbers represent a higher level of satisfaction.
Time Frame: Within 24 hours of the bone marrow sampling procedure
Population: All participants enrolled in the study were included in the analysis as the requires sample size for the study was met. No participants were excluded from analysis. Analysis was made per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
units on a scale | 9 (1.0) | 9.2 (1.0)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Amount of Time Lapsed From Needle to Skin Contact to Bone Marrow Biopsy Specimen Acquisition Using the Manual Device and the Powered Device
Description: measurement of the amount of time required to acquire one bone marrow biopsy specimen. timing starts when the bone marrow aspiration and biopsy needle first contacts the skin and ends when the biopsy specimen has been collected.
Time Frame: at time of the bone marrow sampling procedure
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manual bone marrow aspiration and biopsy procedure | Powered bone marrow aspiration and biopsy procedure
Number analyzed (Participants) | 22 | 22
seconds | 252.4 (95.4) | 224.5 (143.9)
Statistical Analysis 1: Comparison: Manual bone marrow aspiration and biopsy procedure vs Powered bone marrow aspiration and biopsy procedure; Test type: Superiority or Other; p = 0.08, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Participants will be assessed for adverse events for the duration of the bone marrow sampling procedure, an average of 4 hours.
Description: Adverse events reported to the investigators subsequent to a participant's participation will be investigated.
Arm/Group | Manual Bone Marrow Aspiration and Biopsy Procedure | Powered Bone Marrow Aspiration and Biopsy Procedure
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No